CLINICAL TRIAL: NCT05305521
Title: Clinical and Radiographic Outcomes Following Transcrestal Maxillary Sinus Floor Elevation With Injectable Xenogeneic Bone Substitute in Gel Form: a Prospective Multicenter Study
Brief Title: Transcrestal Maxillary Sinus Floor Elevation With Injectable Bone Substitute
Acronym: INJTSFEXEN
Status: Completed | Type: Observational
Sponsor: International Piezosurgery Academy (Other)
Collaborators: Teresa Lombardi DDS private practice (Unknown); Fabio Bernardello MD, DDS private practice (Unknown); Luca Lamazza DDS, PhD private practice (Unknown); Grzegorz Zietek DDS private practice (Unknown); Giuseppe Troiano DDS, PhD private practice (Unknown)
Responsible Party: Principal Investigator, Mr. Claudio Stacchi, DDS, MSc, Claudio Stacchi, DDS, MSc, International Piezosurgery Academy
Other Study IDs: INJTSFE_22
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Edentulous Alveolar Ridge

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Injectable TSFE: partially edentulous patients needing unilateral sinus floor elevation (residual crestal height <5 mm) for the placement of a single implant
  Interventions: Procedure: transcrestal sinus floor elevation; Procedure: Implant placement

INTERVENTIONS:
Procedure: transcrestal sinus floor elevation — Under local anesthesia (articaine 4% with epinephrine 1:100.000), a minimally invasive full-thickness flap was elevated to expose the alveolar crest. Clinicians were left free to choose their preferred transcrestal antrostomy technique. After checking sinus membrane integrity with visual inspection and Valsalva maneuver, pre-heated (40°C) xenogeneic porcine bone substitute in gel form (Gel 40, Tecnoss, Giaveno, Italy) was injected through the crestal antrostomy in order to elevate the membrane and fill the sub-antral space. Duration of graft injection (in seconds) was recorded using a digital chronometer. Periapical intraoperative radiographs were taken to confirm membrane elevation of at least 10 mm.
  Other Names: crestal maxillary sinus lift
Procedure: Implant placement — Simultaneous implant placement was performed when it was possible to achieve adequate primary stability in the residual crestal bone, otherwise crestal antrostomy was sealed by collagen sponges (Hemocollagene, Septodont, Saint-Maur-des-Fossés, France) and implant insertion was postponed.
  Flaps were sutured with Sentineri technique and single stitches using synthetic monofilament
  Other Names: implant insertion

SUMMARY:
To investigate clinical outcomes of transcrestal maxillary sinus floor elevation performed with an injectable xenograft in gel form, analyzing variables possibly influencing the results. Patients needing unilateral sinus floor elevation (residual crestal height <5 mm) for the placement of a single implant were enrolled. Xenograft in gel form was injected through a crestal antrostomy in order to elevate sinus membrane and fill the sub-antral space. Simultaneous implant placement was performed when adequate primary stability was achievable. Graft height was measured immediately after surgery (T0) and after six months of healing (T1). Univariate and multivariate regression models were built to assess associations between clinical variables with implant survival and graft height at T1.

DETAILED DESCRIPTION:
Purpose: To investigate clinical outcomes of transcrestal maxillary sinus floor elevation performed with an injectable xenograft in gel form, analyzing variables possibly influencing the results. Methods: Patients needing unilateral sinus floor elevation (residual crestal height <5 mm) for the placement of a single implant were enrolled. Xenograft in gel form was injected through a crestal antrostomy in order to elevate sinus membrane and fill the sub-antral space. Simultaneous implant placement was performed when adequate primary stability was achievable. Graft height was measured immediately after surgery (T0) and after six months of healing (T1). Univariate and multivariate regression models were built to assess associations between clinical variables with implant survival and graft height at T1.

ELIGIBILITY:
Inclusion Criteria:

* residual bone crest height <5 mm and width ≥6 mm in the planned implant site;
* healed bone crest (at least 6 months elapsed from tooth loss/extraction);
* age >18 years;
* written informed consent given

Exclusion Criteria:

absolute medical contraindications to implant surgery;

* uncontrolled diabetes (HBA1c > 7.5%);
* treated or under treatment with antiresorptives;
* irradiated in the head and neck area in the last five years;
* pregnant or breastfeeding;
* substance abusers;
* psychiatric problems or unrealistic expectations;
* patient not fully able to comply with the study protocol.
* large sinus cavity (distance >12 mm between buccal and palatal walls at 10-mm level, comprising the residual alveolar crest);
* maxillary sinus conditions contraindicating sinus floor elevation;
* poor oral hygiene and motivation (Full Mouth Plaque Score >20% and or Full Mouth Bleeding Score >10%)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any partially edentulous patient needing unilateral sinus floor elevation for the placement of one dental implant supporting a single crown was eligible for entering this study
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
implant survival | 12 months
  implant survival rate after one year of prosthetic loading

SECONDARY OUTCOMES:
vertical bone gain | six months
  vertical bone gain (measured in mm on x-ray) six months after sinus augmentation
percentual graft shrinkage | six months
  % graft shrinkage during 6-month healing period
occurrence of complications | 12 months
  occurrence of any complication or adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Lombardi, Dr., Principal Investigator — International Piezoelectric Surgery Academy
Locations (2):
- Italy (2):
  - Hesire, Cassano Allo Ionio, CS
  - Studio B, Verona, VR

IPD SHARING:
Plan to Share IPD: No
no sharing

REFERENCES:
- [Result] Stacchi C, Spinato S, Lombardi T, Bernardello F, Bertoldi C, Zaffe D, Nevins M. Minimally Invasive Management of Implant-Supported Rehabilitation in the Posterior Maxilla, Part I. Sinus Floor Elevation: Biologic Principles and Materials. Int J Periodontics Restorative Dent. 2020 May/Jun;40(3):e85-e93. doi: 10.11607/prd.4497. PMID 32233183
- [Result] Stacchi C, Spinato S, Lombardi T, Bernardello F, Bertoldi C, Zaffe D, Nevins M. Minimally Invasive Management of Implant-Supported Rehabilitation in the Posterior Maxilla, Part II. Surgical Techniques and Decision Tree. Int J Periodontics Restorative Dent. 2020 May/Jun;40(3):e95-e102. doi: 10.11607/prd.4498. PMID 32233185
- [Derived] Lombardi T, Lamazza L, Bernardello F, Zietek G, Stacchi C, Troiano G. Clinical and radiographic outcomes following transcrestal maxillary sinus floor elevation with injectable xenogenous bone substitute in gel form: a prospective multicenter study. Int J Implant Dent. 2022 Jul 22;8(1):32. doi: 10.1186/s40729-022-00431-5. PMID 35867239